CLINICAL TRIAL: NCT00606710
Title: Cognis and Teligen 100 HE and Reliance Quadripolar Defibrillation Lead (4-Site) Field Following
Acronym: Cogent-4
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Torsten Kayser, Boston Scientific
Other Study IDs: Cogent-4 0806
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Ventricular Tachycardia, Ventricular Fibrillation; Heart Failure
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cognis 100-D, Teligen DR, VR 100 HE — ICD or CRT - Therapy
  Other Names: Reliance Quadripolar Defibrillation Lead

SUMMARY:
The COGENT-4 Field Following Study will evaluate the clinical performance of the Boston Scientific TELIGEN 100 HE Implantable Cardioverter Defibrillator (ICD), the COGNIS 100 HE Cardiac Resynchronization Therapy ICD (CRT-D) systems and the RELIANCE 4-SITE defibrillation lead (when available). An optional sub-study will also evaluate the clinical performance of the Reverse Mode Switch (RMS) feature in the TELIGEN 100 HE DR ICD.

ELIGIBILITY:
Inclusion Criteria:

* ICD indication according to normal clinical practice (for those patients receiving a TELIGEN 100 HE)
* CRT-D indication according to normal clinical practice (for those patients receiving a COGNIS 100 HE)
* Willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigational centre and at the intervals defined by this protocol
* Geographically stable patients who are available for follow-up at a study centre
* Age 18 or above, or of legal age to give informed consent specific to national law

Exclusion Criteria:

* Documented life expectancy of less than six months or expected to undergo heart transplant within the next six months
* Patients currently requiring dialysis
* Women who are pregnant or plan to become pregnant. Method of assessment per physician discretion
* Enrolled in any concurrent study
* Patients implanted with the following leads which will not be abandoned:
* Atrial or right ventricular unipolar leads
* Patch defibrillation leads
* Non-compatible defibrillation leads (e.g. 5/6mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with risk of developing life threatening ventricular arrhythmias with and without heart failure
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Appropriate detection of ventricular arrhythmias | Predischarge

SECONDARY OUTCOMES:
Appropriate shock conversion | Predischarge

CONTACTS AND LOCATIONS:
Overall Officials: Poul Erik Bloch Thomsen, MD, Principal Investigator — KAS Gentofte Hospital
Locations (4):
- KAS Gentofte Hospital, Hellerup, Denmark
- Israel (3):
  - Barzilay Medical Center, Ashkelon
  - Tel Aviv Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky